CLINICAL TRIAL: NCT03527940
Title: Prognostic Markers of Patients With ST-segment Elevation Myocardial Infarction
Brief Title: Prognostic Markers of Patients With STEMI
Status: Completed | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, Dr, Chongqing Medical University
Other Study IDs: 2018-32-1
Record Dates: First submitted 2018-05-05; First posted 2018-05-17 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with STEMI

SUMMARY:
To analyze the relationship between the clinical data and the outcomes of STEMI patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ST-segment elevation myocardial infarction(STEMI).

Exclusion Criteria:

* Patients with concurrent infection or any documented inflammatory illness, such as arthritis or connective tissue diseases,or any other malignancy.
* Pregnant women.
* Severe hepatic dysfunction.
* Uncontrolled hypertension.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with STEMI
Sampling Method: Non-Probability Sample
Enrollment: 932 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dongying Zhang, PhD, Study Director — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China